CLINICAL TRIAL: NCT06146413
Title: Triggering Oocyte Maturation in Normoresponders Using Double Trigger or HCG Trigger . A Randomized Controlled Trial
Brief Title: Triggering Oocyte Maturation in Normoresponders Using Double Trigger or HCG Trigger
Acronym: Doubtrig
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bedaya Hospital (Other)
Responsible Party: Principal Investigator, Usama M.Fouda, Clinical Professor, Bedaya Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Double trigger in IVF
Record Dates: First submitted 2023-11-19; First posted 2023-11-24 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Infertility
Keywords: Infertility; IVF-ET; HCG trigger; Double trigger
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Double trigger (Experimental): GnRH agonist ( Triptorelin ) ( 0.2 mg / S.C ) and hCG ( 10000 IU) are administered 40 and 34 h before oocyte retrieval
  Interventions: Drug: Double trigger
- HCG trigger (Active Comparator): HCG ( 100000 IU/ I.M ) is administered 36 h before oocyte retrieval
  Interventions: Drug: HCG trigger

INTERVENTIONS:
Drug: Double trigger — GnRH agonist ( Triptorelin ) ( 0.2 mg / S.C ) and hCG ( 10000 IU) are administered 40 and 34 h before ovum pick-up
  Other Names: Augmented trigger
  Arms: Double trigger
Drug: HCG trigger — hCG ( 10000 IU) is administered 36 h before ovum pick-up
  Other Names: Conventional trigger
  Arms: HCG trigger

SUMMARY:
The aim of this study is to compare the efficacy double trigger [ co-administration of GnRH agonist with HCG 40 and 34 h prior to ovum pick-up, respectively] with HCG trigger in inducing oocyte maturation.

DETAILED DESCRIPTION:
Several studies revealed that the double trigger regimen was effective in the treatment of patients with a history of immature oocytes retrieved or with suboptimal oocytes yield.

The investigators designed this randomized controlled trial to compare the efficacy double trigger with HCG trigger in inducing oocyte maturation.in normoreponders undergoing IVF-ET

ELIGIBILITY:
Inclusion Criteria:

* Normoresponders
* GnRH antagonist cycles

Exclusion Criteria:

* BMI more than 35
* Endometriosis
* AMH less than 1.1 ng
* AMH more than 4
* PCOS
* Poor responders

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 150 (Estimated)
Dates: Start 2023-12-30 (Estimated); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Metaphase-II oocytes rate | Ten to fifteen days after starting ovarian stimulation
  Number of MII oocyte/ number of cumulus oocyte complex

SECONDARY OUTCOMES:
Clinical pregnancy rate | 5 weeks after embryo transfer
  Presence of intrauterine gestational sac detected by transvaginal ultrasound
Ongoing Pregnancy Rate | 18 weeks after embryo transfer
  Pregnancies continued beyond 20 weeks gestation

CONTACTS AND LOCATIONS:
Overall Officials: Ismail Aboul Foutouh, Prof., Study Chair — Cairo University
Locations (1):
- Bedaya Hospital, Giza, Egypt

REFERENCES:
- [Background] Haas J, Zilberberg E, Dar S, Kedem A, Machtinger R, Orvieto R. Co-administration of GnRH-agonist and hCG for final oocyte maturation (double trigger) in patients with low number of oocytes retrieved per number of preovulatory follicles--a preliminary report. J Ovarian Res. 2014 Aug 2;7:77. doi: 10.1186/1757-2215-7-77. PMID 25296696